CLINICAL TRIAL: NCT00353418
Title: A Randomized, Multicenter, Double Blinded Study Comparing the Safety and Efficacy of Pegasys® 180 ug Plus Copegus® 1000 or 1200 mg to the Currently Approved Combination of Pegasys® 180 ug Plus Copegus® 800 mg in Interferon-naïve Patients With Chronic Hepatitis C Genotype 1 Virus Infection and HIV-1
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) Plus COPEGUS (Ribavirin) in Patients With Chronic Hepatitis C (CHC) Genotype 1 and Human Immunodeficiency Virus-1 (HIV-1) Co-infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV18209
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Results first posted 2010-06-15 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg (Experimental)
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg (Active Comparator)
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 180 µg subcutaneously weekly for 48 weeks
  Other Names: Pegasys
Drug: Ribavirin — 800 mg orally daily for 48 weeks
  Other Names: Copegus
  Arms: PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg
Drug: Ribavirin — 1000 mg or 1200 mg (based on patient weight of < 75 kg or ≥ 75 kg, respectively) orally daily for 48 weeks
  Other Names: Copegus
  Arms: PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg

SUMMARY:
This 2-arm study will compare the efficacy and safety of treatment with Pegasys (180 µg weekly) plus Copegus (800 mg daily) and Pegasys (180 µg weekly) plus Copegus (1000-1200 mg daily) in interferon-naive patients with CHC genotype 1 co-infected with HIV-1. Treatment will be administered for 48 weeks, and this will be followed by 24 treatment-free weeks. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥18 years of age
* CHC genotype 1
* Stable HIV-1 infection

Exclusion Criteria:

* Previous treatment with an alpha interferon, ribavirin, viramidine, levovirin, amantadine or investigational HCV protease or polymerase inhibitors
* Medical condition associated with liver disease other than CHC infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

REFERENCES:
- [Derived] Rodriguez-Torres M, Slim J, Bhatti L, Sterling R, Sulkowski M, Hassanein T, Serrao R, Sola R, Bertasso A, Passe And S, Stancic S. Peginterferon alfa-2a plus ribavirin for HIV-HCV genotype 1 coinfected patients: a randomized international trial. HIV Clin Trials. 2012 May-Jun;13(3):142-52. doi: 10.1310/hct1303-142. PMID 22592094

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg
Started | 138 | 277
Completed | 55 | 119
Not Completed | 83 | 158

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg | Total
Number analyzed (Participants) | 138 | 277 | 415
Age, Customized [Number; unit: Participants] — The All Patients Treated population included all patients randomized who had received at least one dose of study medication: PEG-IFN alfa 2-a 180 μg + ribavirin 800 mg = 135 patients; PEG-IFN alfa 2-a 180 μg + ribavirin 1000 or 1200 mg = 275 patients.
  Participants
    < 65 years | 134 | 273 | 407
    >=65 years | 1 | 2 | 3
Age Continuous [Mean (Standard Deviation); unit: Years] — The All Patients Treated population included all patients randomized who had received at least one dose of study medication: PEG-IFN alfa 2-a 180 μg + ribavirin 800 mg = 135 patients; PEG-IFN alfa 2-a 180 μg + ribavirin 1000 or 1200 mg = 275 patients.
  Years | 45.2 (8.39) | 45.5 (8.16) | 45.4 (8.24)
Gender [Number; unit: Participants] — The All Patients Treated population included all patients randomized who had received at least one dose of study medication: PEG-IFN alfa 2-a 180 μg + ribavirin 800 mg = 135 patients; PEG-IFN alfa 2-a 180 μg + ribavirin 1000 or 1200 mg = 275 patients.
  Participants
    Female | 29 | 51 | 80
    Male | 106 | 224 | 330

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response (SVR)
Description: SVR was defined by the percentage of patients with undetectable Hepatitis C virus (HCV) ribonucleic acid (RNA) at 24 weeks after completion of the 48-week treatment period (i.e., a single last HCV RNA < 20 IU/mL measured ≥ Day 477 [≥ Week 68]). Patients without an HCV measurement at the end of the 24-week untreated follow-up period were considered nonresponders.
Time Frame: Week 72
Population: The All Patients Treated population included all patients randomized who had received at least one dose of study medication: PEG-IFN alfa 2-a 180 μg + ribavirin 800 mg = 135 patients; PEG-IFN alfa 2-a 180 μg + ribavirin 1000 or 1200 mg = 275 patients.
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg
Number analyzed (Participants) | 135 | 275
Percentage of participants | 19 | 22
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg vs PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg; Sample sizes of 133 and 267 patients for RBV 800 mg daily and RBV 1000 or 1200 mg daily, respectively, provided the following probabilities of detecting the specified differences in SVR with a 0.05 level two-sided chi-square test of significance: RBV 800 mg SVR - 0.30; RBV 1000 or 1200 mg SVR - 0.40; Probability - 0.49 RBV 800 mg SVR - 0.30; RBV 1000 or 1200 mg SVR - 0.45; Probability - 0.83; Test type: Superiority or Other; p = 0.6119, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.15, 95% CI [0.68 to 1.93]

2. Secondary Outcome: Virological Response at End of Treatment Period
Description: Virological response at the end of the treatment period was defined as a single last HCV RNA measurement <20 IU/mL at the completion of the treatment period (Days 324 to 351). Patients without an HCV measurement at Week 48 were considered nonresponders.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg
Number analyzed (Participants) | 135 | 275
Percentage of participants | 30 | 35

3. Secondary Outcome: Virological Response at Weeks 4, 12 and 24
Description: Virological response at Weeks 4, 12 and 24 was also defined as a single last undetectable HCV RNA (< 20 IU/mL) falling within the visit windows of Days 16 to 43, 72 to 99, and 156 to 183, respectively. Patients without an HCV measurement at a study week were considered nonresponders at that study week.
Time Frame: Weeks 4, 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg
Number analyzed (Participants) | 135 | 275
Percentage of participants
  Week 4 | 8 | 7
  Week 12 | 25 | 25
  Week 24 | 33 | 40

4. Secondary Outcome: Relapse of Virological Response
Description: Relapse of virological response was calculated by dividing the number of patients who achieved a virological response at the end of treatment but had detectable HCV RNA at the last assessment posttreatment by the number of patients with a virological response at the end of treatment who had at least one HCV RNA assessment posttreatment.
Time Frame: Weeks 48 and 72
Population: Within the All Patients Treated population, patients with a response at end of treatment: PEG-IFN alfa 2-a 180 μg + ribavirin 800 mg = 37 patients; PEG-IFN alfa 2-a 180 μg + ribavirin 1000 or 1200 mg = 83 patients.
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg
Number analyzed (Participants) | 37 | 83
Percentage of participants | 32 | 36

5. Secondary Outcome: Rapid Virological Response (RVR) by Week 4
Description: RVR was defined as an undetectable HCV RNA < 20 IU/mL (a single last HCV RNA < 20 IU/mL falling in the time window of Days 2 to 43). Patients without an HCV measurement by Week 4 were considered nonresponders.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg
Number analyzed (Participants) | 135 | 275
Percentage of participants | 8 | 7

6. Secondary Outcome: Early Virological Response (EVR), Partial EVR and Complete EVR by Week 12
Description: EVR: Undetectable HCV RNA <20 IU/mL or ≥2 log10 drop from pretreatment level, by Week 12 (a single last HCV RNA <20 IU/mL or ≥2 log10 drop from pretreatment level in the time window of Days 2 to 99). Partial EVR: Detectable HCV RNA but ≥2 log10 drop from pretreatment, by Week 12 (a single last HCV RNA detectable but ≥2 log10 drop from pretreatment in the time window of Days 2 to 99). Complete EVR: Undetectable HCV RNA <20 IU/mL, by Week 12 (a single last HCV RNA <20 IU/mL in the time window of Days 2 to 99). Patients without an HCV measurement by Week 12 were considered nonresponders.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg
Number analyzed (Participants) | 135 | 275
Percentage of participants
  Early Virological Response | 51 | 61
  Partial Early Virological Response | 25 | 35
  Complete Early Virological Response | 26 | 26

7. Primary Outcome: Incidence of Adverse Events, Dose Reductions and Withdrawals Due to Anemia
Description: Adverse events of anemia included hemolytic anemia, aplasia pure red cell, and pancytopenia.
Time Frame: Up to Week 72
Population: The Safety population included all patients randomized who received at least one dose of the study medication and had at least one postbaseline safety assessment: PEG-IFN alfa 2-a 180 μg + ribavirin 800 mg = 135 patients; PEG-IFN alfa 2-a 180 μg + ribavirin 1000 or 1200 mg = 274 patients.
Measure: Number; unit: Percentage of participants
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg
Number analyzed (Participants) | 135 | 274
Percentage of participants
  Adverse anemic event | 24 | 32
  Serious adverse anemic event | 4 | 4
  PEG-INF alfa-2a dose modification due to anemia | 2 | 3
  Ribavirin dose modification due to anemia | 10 | 18
  Premature PEG-INF alfa-2a withdrawal due to anemia | 1 | 3
  Premature ribavirin withdrawal due to anemia | 2 | 3

ADVERSE EVENTS:
Description: The Safety population included all patients randomized who received at least one dose of the study medication and had at least one postbaseline safety assessment: PEG-IFN alfa 2-a 180 μg + ribavirin 800 mg = 135 patients; PEG-IFN alfa 2-a 180 μg + ribavirin 1000 or 1200 mg = 274 patients.
Arm/Group | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg
Serious Adverse Events (participants affected / at risk) | 21/135 | 46/274
Other Adverse Events (participants affected / at risk) | 132/135 | 264/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg (N=135) | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg (N=274)
Bronchitis (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia Pneumococcal (Infections and infestations) | 1 | 1
Staphylococcal Abscess (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2
Anal Abscess (Infections and infestations) | 0 | 1
Bursitis Infective (Infections and infestations) | 0 | 1
Carbuncle (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumococcal Bacteraemia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Subdiaphragmatic Abscess (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 8
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Autoimmune Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 2
Completed Suicide (Psychiatric disorders) | 0 | 1
Substance Abuse (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Hypertrophic Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 1
Splenic Injury (Injury, poisoning and procedural complications) | 0 | 1
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain Stem Ischaemia (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Optic Neuritis (Nervous system disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a 180 μg + Ribavirin 800 mg (N=135) | PEG-IFN Alfa-2a 180 μg + Ribavirin 1000 or 1200 mg (N=274)
Fatigue (General disorders) | 64 | 129
Pyrexia (General disorders) | 36 | 63
Chills (General disorders) | 26 | 44
Irritability (General disorders) | 20 | 32
Pain (General disorders) | 14 | 32
Asthenia (General disorders) | 14 | 29
Malaise (General disorders) | 8 | 18
Nausea (Gastrointestinal disorders) | 35 | 69
Diarrhoea (Gastrointestinal disorders) | 31 | 60
Vomiting (Gastrointestinal disorders) | 20 | 25
Abdominal Pain (Gastrointestinal disorders) | 8 | 13
Dyspepsia (Gastrointestinal disorders) | 4 | 17
Constipation (Gastrointestinal disorders) | 7 | 10
Insomnia (Psychiatric disorders) | 35 | 78
Anxiety (Psychiatric disorders) | 16 | 26
Headache (Nervous system disorders) | 48 | 93
Dizziness (Nervous system disorders) | 17 | 30
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 27
Urinary Tract Infection (Infections and infestations) | 5 | 16
Bronchitis (Infections and infestations) | 9 | 10
Anaemia (Blood and lymphatic system disorders) | 33 | 89
Neutropenia (Blood and lymphatic system disorders) | 32 | 62
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 38
Back Pain (Musculoskeletal and connective tissue disorders) | 16 | 19
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 8 | 9
Rash (Skin and subcutaneous tissue disorders) | 12 | 26
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 19
Dry Skin (Skin and subcutaneous tissue disorders) | 9 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 21
Night Sweats (Skin and subcutaneous tissue disorders) | 7 | 10
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 25
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 14
Decreased Appetite (Metabolism and nutrition disorders) | 34 | 61
Weight Decreased (Investigations) | 21 | 50
Depression (Psychiatric disorders) | 30 | 68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.